CLINICAL TRIAL: NCT06836960
Title: The Clinical Efficacy of Gegen Qinlian Tang Combined with Bifidobacterium Triple Viable Capsules in the Prevention and Treatment of Radiation Enteritis
Brief Title: Gegen Qinlian Tang and Probiotics for Radiation Enteritis
Acronym: GQBT-RE
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiujiang No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Lu Wang, Jiujiang NO.1 Hospital, Jiujiang No.1 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JJSDYRMYY-YXLL-2014-193; S2021ZDYFN148 (Other Grant/Funding Number: Jiujiang City Key Research and Development Plan)
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Radiation Enteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Probiotics With Gegen Qinlian Tang Group (Experimental): Participants in this group will receive an oral placebo matched in appearance to the Bifidobacterium Triple Viable Capsules, taken three times daily for 8 weeks. No active interventions will be administered in this group, serving as the placebo control.
  Interventions: Drug: Probiotic Therapy With Gegen Qinlian Tang

INTERVENTIONS:
Drug: Probiotic Therapy With Gegen Qinlian Tang — This intervention includes the oral administration of Bifidobacterium Triple Viable Capsules (0.5 g, three times daily) combined with Gegen Qinlian Tang (200 mL, twice daily) for 8 weeks. The combination therapy is designed specifically for the prevention and treatment of radiation enteritis, differentiating it from probiotics or herbal therapies used alone.

SUMMARY:
The purpose of this clinical study is to evaluate whether Bifidobacterium Triple Viable Capsules, alone or in combination with Gegen Qinlian Decoction, can effectively prevent and treat acute radiation enteritis in patients undergoing abdominal or pelvic radiotherapy.

The study aims to answer the following question: Can probiotics, with or without the addition of herbal medicine, reduce the incidence and severity of radiation-induced intestinal injury and improve the quality of life for patients during and after radiotherapy?

A total of 60 patients with malignant tumors receiving abdominal or pelvic radiotherapy will be recruited and randomly assigned to one of three groups: a control group (no intervention), a probiotics-only group (Bifidobacterium Triple Viable Capsules, three capsules twice daily), and a combination therapy group (probiotics with modified Gegen Qinlian Decoction tailored to individual symptoms).

The primary outcome will be the incidence and severity of acute radiation enteritis, assessed using the RTOG/EORTC grading criteria (0-IV levels). Daily observations will be recorded during radiotherapy, with follow-up lasting three months after the completion of treatment.

This study seeks to provide evidence for the use of probiotics and herbal medicine as effective strategies to mitigate the side effects of radiotherapy and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:1.Age:Participants aged 18 to 80 years.2.Diagnosis:

Patients diagnosed with malignant tumors confirmed by cytological or pathological examination.Patients scheduled for abdominal or pelvic radiotherapy based on treatment guidelines.3Cognitive and Communication Ability:Participants must have clear consciousness and normal cognitive abilities to communicate effectively.4.Consent:Participants must provide written informed consent and agree to participate in the study.

Family members must also provide consent if applicable.5.Willingness to Cooperate:Participants must be willing to comply with the study procedures and requirements.

Exclusion Criteria:1.History of Severe Intestinal Diseases:Patients with a history of severe intestinal diseases, including ischemic bowel disease, ulcerative colitis, Crohn's disease, or other chronic inflammatory bowel conditions.2.Recent Antibiotic Use:Patients who have received antibiotic treatment within the past 2 years.3.Severe Organ Dysfunction:Patients with severe liver or kidney dysfunction, as determined by clinical assessment or laboratory tests.4.Comorbidities and Other Major Diseases:

Patients with other serious illnesses that may interfere with the study protocol or compliance, including but not limited to cardiovascular, respiratory, or neurological diseases.5.Inability to Participate:Patients unable to cooperate with the study procedures due to physical or psychological reasons.Patients who are likely to withdraw midway through the study.6.Incomplete Medical Records or Refusal to Share Data:Patients who refuse to share their medical records or have incomplete medical documentation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Radiation Enteritis | From the start of radiotherapy to 3 months post-treatment
  The incidence of acute radiation enteritis will be assessed using the RTOG/EORTC grading criteria (Grade 0-IV). Symptoms such as diarrhea, abdominal pain, and mucus secretion will be monitored daily during radiotherapy and up to three months post-treatment. The outcome will measure the proportion of patients experiencing Grade II or higher symptoms in each study arm. This assessment aims to evaluate the effectiveness of Bifidobacterium Triple Viable Capsules, alone or in combination with Gegen Qinlian Decoction, in reducing the incidence of radiation enteritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiujiang NO.1 People's Hospital, Jiujiang, Jiangxi, China